CLINICAL TRIAL: NCT05828251
Title: Full Thickness Macular Hole; Should it be Handled Subacutely?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Asrin Rasul, Medical Doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rigshospitalet-RS studie
Record Dates: First submitted 2023-03-22; First posted 2023-04-25 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Full Thickness Macular Hole
Keywords: Phako; Vitrectomy; Phako-vitrectomy; FTMH
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in the first part om of the study, 28 patients in each arm.
  Prospective study in second part of the study with 28 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Phako-Vitrectomy for FTMH (Experimental): Study 1: Patient randomized to this arm will receive a combined phako-vitrectomy within two weeks from referall day.
  Interventions: Procedure: Combined phako-vitrectomy
- Sequential phako and vitrectomy for FTMH (Active Comparator): Study 1: Patients randomized to this arm will receive a standard phacoemulsification as soon as possible. About four weeks after phacoemulsification a vitrectomy is performed.
  Interventions: Procedure: Vitrectomy (Sequential phakoemulsification and vitrectomy); Procedure: Phako (Sequential phakoemulsification and vitrectomy)
- Longstanding FTMH (Other): Study 2: Patients with symptomduration of 3-12 months will be included in this part of the study in a prospective design.
  Interventions: Procedure: Vitrectomy (Sequential phakoemulsification and vitrectomy); Procedure: Phako (Sequential phakoemulsification and vitrectomy)

INTERVENTIONS:
Procedure: Vitrectomy (Sequential phakoemulsification and vitrectomy) — Standard treatment for FTMH at our department with phakoemulsification followed by pars plana vitrectomy and gas 4 weeks later.
  Arms: Longstanding FTMH; Sequential phako and vitrectomy for FTMH
Procedure: Combined phako-vitrectomy — Phakoemulsication and pars plana vitrectomy are performed in the same setting. This procedure is normally only offeres to selected cases at our department.
  Arms: Combined Phako-Vitrectomy for FTMH
Procedure: Phako (Sequential phakoemulsification and vitrectomy) — Standard treatment for FTMH at our department with phakoemulsification followed by pars plana vitrectomy and gas 4 weeks later.
  Arms: Longstanding FTMH; Sequential phako and vitrectomy for FTMH

SUMMARY:
Full thickness macular hole, FTMH, is a retinal disease involving the fovea that cause central vision loss, metamorphopsia and central scotoma. The most effective treatment for FTMH is a pars plana vitrectomy and a tamponade with expansile gas. It is well known that vitrectomy accelerates cataract development. Vitrectomy can therefore be combined with cataract surgery in the same setting, a procedure that is shown to be safe, although increased inflammation and rates of central macular edema have been reported in some studies. Cataract surgery can also be performed prior or deferred until compromising the visual acuity after vitrectomy. Cataract-surgeries are more challenging in vitrectomized eyes due to lack of vitreous support and risk of loose zonules. The normal practice for FTMH at our department is therefore cataract surgery followed by vitrectomy 4 weeks later. A combined phaco-vitrectomy procedure is offered to patients who are at the labor market or when general anesthesia is required for the surgery. In non-presbyopic patients (<50 years) only vitrectomy is performed.

The visual improvement after surgery seems to be dependent on preoperative characteristics, such as the preoperative visual acuity, size of the hole and the duration of symptoms. The duration of symptoms is a known prognostic factor, and recently shown that the longer duration, the worse visual outcome. The precise timeframe for the optimal final outcome is not known.

The combined surgery is known to be safe in the treatment for epiretinal membrane, where a intravitreal gasfill is not necessary. However, the use of gas in FTHM surgery causes risk of increased movement of the newly inserted intraocular lens. This can lead to increased anterior segment inflammation with ensuing vision threatening cystic macular edema, as mentioned above.

The purpose of this study is to investigate whether small FTMH with a short duration of symptoms have better visual outcome with a prompt combined phako-vitrectomy (within two weeks), compared to the current standard of care of receiving cataract surgery as soon as possible and vitrectomy 4 weeks later. How the delay of surgery affects the visual outcome will also be investigated, by including patients with longer duration of symptoms. The main hypothesis is that the chance of better visual outcome is higher for macular holes with early surgery compared to the current standard of care and that the duration of symptoms has significant impact on the visual outcome.

Method

The study consists of 2 parts.

1. Patients with idiopathic FTMH <400µm in diameter (as defined by The international vitreomacular traction study group classification), with a duration of symptoms of less than 30 days will be randomized into 2 groups:

   Group1: Combined phaco-vitrectomy within 2 weeks (after referral). Group 2: Current standard of care with cataract surgery as soon as possible and vitrectomy 4 weeks later.
2. Group 3: Patients with small holes <400µm, with a duration of symptoms of more than 3 months and less than one year will be included in this part of the study. These patients will be treated and followed as in Group 2.

They will be reviewed a total of 7 times in Group 1 and 9 times in Group 2 and 3: a preoperative examination followed by 6/8 postoperative examinations. Additional examinations will be scheduled if needed.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic full thickness macular hole
* Duration of symptoms of <30 days for Group 1 and 2
* Duration of symptoms of 3-12 months for Group 3
* FTMH size <400µm
* >18 years
* Able to give informed consent
* Compliance for postoperative positioning

Exclusion Criteria:

* High myopia (≤-3)
* Traumatic macular hole
* Prior ocular surgery, including cataract surgery
* Other ocular diseases compromising the visual acuity (i.e., AMD, diabetic retinopathy, previous vein occlusion)
* Posterior vitreous detachment (Weiss ring)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 12 months after vitrectomy
  Best corrected visual acuity measured with ETDRS, the ETDRS scoe will be converted to LogMAR

SECONDARY OUTCOMES:
Metamorphopsia | 12 months after vitrectomy
  Measured by M-charts, for vertical and horisontal metamorfopisa. The M-charts consist of 19 dotted (dot size is 0.1°) lines with dot intervals ranging from 0.2° to 2.0° of visual angle.
Hole closure rates | Measured 4 weeks after surgery
  Either the hole closes og it doesn't.
Microperimetry | 12 months after surgery
  Microperimetry is a procedure to assess retinal sensitivity while fundus is directly examined; it enables exact correlation between macular pathology and corresponding functional abnormality. Measured in mean retinal sensitivity (dB)
Anterior chamber inflammation | 1 day and 1 week after the first surgery
  (FM). The FM is based on the measurement principle of laser light scattering detection. The instrument uses a diode laser beam to scan a measuring window that is projected inside the anterior chamber of the eye. As an aqueous protein (component of inflammation) passes through the focal point of the laser,light scattering occurs. The intensity of the scattered light (directly proportional to the amount of protein particles-flare) is detected by a photo-multiplier tube (PMT), which generates an electrical signal. This signal is immediately digitized to eliminate outside noise interference and are processed by a computer which displays the results for user analysis. The unit of measurement employed by the FM is "Photon Count" per millisecond.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Dornonville de la Cour, MD, Prof., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Denmark, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No